CLINICAL TRIAL: NCT01958931
Title: Evaluate the Utility of the ProLung Test as Adjunctive to CT Scan in the Diagnosis of Lung Cancer
Status: Completed | Type: Observational
Sponsor: Fresh Medical Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: FML - 204
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Solitary Pulmonary Nodule; Multiple Pulmonary Nodules
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients Suspicious for Lung Cancer: Subjects are symptomatic of lung cancer and have one or more lung nodules or lung masses suspicious for lung cancer.

SUMMARY:
A Study to evaluate the utility of the ProLung Test as an adjunct to CT scan in the diagnosis of lung cancer.

DETAILED DESCRIPTION:
This Study will assess the stability of the ProLung Test classification algorithm when used as an adjunct to CT scan. This Study will assess whether there are any potential safety concerns of the ProLung Test when used to evaluate patients with a positive CT scan for lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, age 18 or above.
* If female, subject

  * is of non-childbearing potential meaning permanently sterile, or
  * is one year post-menopausal; or
  * is not pregnant as confirmed by negative urine pregnancy test and using adequate birth control at time of screening.
* Subject presents with one or more of the following clinical symptoms or suspicious radiological finding(s):

  * Persistent cough
  * Hoarseness
  * Shortness of breath
  * Sputum streaked with blood
  * Fatigue
  * Unexplained recent weight loss
  * Recurrent pneumonia or bronchitis
  * Chest pain
  * Abnormal chest radiograph
* Subject has undergone a CT scan of the lungs within 44 days of measurement that indicates one or more non-calcified nodules (NCN) or lung masses suspicious for lung cancer.
* Subject is capable of understanding and agreeing to fulfill the requirements of this protocol.
* Subject has signed the IRB/IEC approved informed consent form.

Exclusion Criteria:

• Subjects who meet one or more of the following criteria may not be enrolled in this Study:

* Subject has a pacemaker or other implanted electronic device.
* Subject with diagnosed malignancy within the past 5 (five) years except for non-melanoma skin cancer.
* Subject with significant systemic diseases including uncontrolled diabetes, severe heart failure, uncontrolled hypertension, myocardial infarction and/or auto-immune conditions within the prior 3 (three) months.
* Subject taking systemic corticosteroid medication (except for inhaled) within 14 days prior to measurement session.
* Subject has had an invasive medical procedure that involves the thoracic cavity within 30 days prior to the measurement session.
* Subject who currently abuses alcohol or drugs.
* Subject presents with an anomalous physical or anatomical condition that precludes measurement.
* Subject will have undergone unusually strenuous exercise within 24 hours prior to measurement session.
* Subject who has, in the Principal Investigator's opinion, any medical condition or other circumstance that would prevent completion of this Study or interfere with analysis of the Study results.
* Subjects who have undergone radiation and chemotherapy treatment within the past 30 days.
* Subject receiving therapy for documented or suspected chest infection.
* Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with lung cancer symptoms and pulmonary lesions suspicious for lung cancer
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2007-09; Primary Completion 2008-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
ProLung Test utility in lung cancer | date of conclusive diagnosis
  This Study will assess the stability of the ProLung Test classification algorithm when used as an adjunct to CT scan to determine whether it is appropriate to be used in a pivotal study.

SECONDARY OUTCOMES:
Safety and Tolerability of the ProLung Test | within 30 minutes of the ProLung Test
  This Study will assess whether there are any potential safety concerns of the ProLung Test when used to evaluate patients with a positive CT scan for lung cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States